CLINICAL TRIAL: NCT00653341
Title: Target Glycemic Control and the Incidence of Symptomatic Nocturnal Hypoglycemia in Insulin Naïve Subjects With Type 2 Diabetes on Oral Hypoglycemic Agent(s) and Treated With Insulin Glargine or NPH Human Insulin.
Brief Title: Effect of Insulin Glargine in Insulin Naïve Subjects With Type 2 Diabetes on Oral Hypoglycemic Agent(s)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, Sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901/4002
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: insulin naive
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin, Isophane

INTERVENTIONS:
Drug: insulin glargine
Drug: NPH human insulin

SUMMARY:
The primary objective of this study is to compare the percentage of subjects who reach the target HbA1c level (< or = 7.0% at endpoint) and do not experience symptomatic nocturnal hypoglycemia during treatment with insulin glargine or NPH human insulin.

ELIGIBILITY:
Inclusion Criteria:

* Insulin naïve subjects with type 2 diabetes treated with oral hypoglycemic agents
* Body mass index between 26 and 40 kg/m2
* HbA1c between 7.5% and 10.0%
* Fasting plasma glucose >7.8 mmol/L and fasting C-peptide > or =0.25 nmol/L

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Actual)
Dates: Start 2000-01; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects reaching target HbA1c = or < 7% at endpoint and not experiencing symptomatic nocturnal hypoglycemia

SECONDARY OUTCOMES:
Safety data (Adverse events, vital signs, laboratory values, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Public Registry ICD, Study Director — Sanofi
Locations (2):
- Sanofi-aventis administrative office, Bridgewater, New Jersey, United States
- Sanofi-aventis administrative office, Laval, Canada

REFERENCES:
- [Result] Riddle MC, Rosenstock J, Gerich J; Insulin Glargine 4002 Study Investigators. The treat-to-target trial: randomized addition of glargine or human NPH insulin to oral therapy of type 2 diabetic patients. Diabetes Care. 2003 Nov;26(11):3080-6. doi: 10.2337/diacare.26.11.3080. PMID 14578243
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419